CLINICAL TRIAL: NCT02517762
Title: Labour Triggered Acute Low Back Pain: Origin, Mechanisms, Causes of Pain, Evaluation of Treatment and Followup
Brief Title: Acute Low Back Pain: Causes, Mechanisms, Treatment and Followup
Acronym: ALBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XC90-ALBP
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Acute Low Back Pain; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stay active (Experimental): Receive the advice by the physician to stay as active as possible in spite of the pain experienced
  Interventions: Behavioral: Physical activity
- Adjust activity (Experimental): Receive the advice by the physician to adjust the activity according to the pain, i.e. to avoid activities, movements or positions that cause or worsen the pain
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity

SUMMARY:
The purpose of this study is to investigate acute low back pain, its origin, mechanisms, the cause of pain, evaluation of treatments and development. Employees from a large local manufacturing company are sent for a complete orthopedic and pain evaluation immediately after onset of acute low back pain. Thereafter, the included patients are allocated either to the advice to stay as active as possible in spite of the pain or to adjust their activity to the pain. Pain intensity and physical activity are followed prospectively over seven days using a diary and a pedometer.

DETAILED DESCRIPTION:
The purpose of this study is to investigate acute low back pain, its origin, mechanisms, the cause of pain, evaluation of treatments and development. Employees from a large local manufacturing company are sent for a complete orthopedic and pain evaluation immediately after onset of acute low back pain. The patients go through x-ray examinations, physical examinations, they complete a battery of questionnaires covering history of acute low back pain, lifestyle characteristics, work place factors, psychosocial factors, and indicate pain intensity and pain locations. Thereafter the patients are randomly allocated to one of two treatment advices: stay active as much as possible in spite of pain or adjust the activity to the pain. During seven days after the medical examination the patients wear a pedometer attached to the waist and annotate the number of steps and pain intensity, pain location and pain-related disability in a diary. A numeric graphic scale is used for pain intensity. Work absenteeism and sick leave due to the current acute back pain is collected from the company records. Immediate inclusion after pain onset is facilitated with continuous communication with the manufactory company. Physical activity and pain development over the seven days is investigated statistically using linear mixed models for repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Severe acute low back pain, duration within 24h after onset, pain exceeds 50mm on the visual analog scale (VAS)

Exclusion Criteria:

* Sick-leave because of low back pain or in spine in the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2005-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Acute low back pain | 7 days
  Pain intensity is assessed from a numerical graphic scale, ranging from 0 (no pain) to 10 (pain as bad as it can be); the patients complete the scale each day in a diary
Physical activity | 7 days
  The patients wear a pedometer attached to the hip and annotate the number of daily steps each day in a diary

SECONDARY OUTCOMES:
Work absenteeism and sick leave | 7 days
  Work absenteeism and sick leave due to the current backpain is collected from the manufacturing company records up to one month after the onset of the acute low back pain

CONTACTS AND LOCATIONS:
Overall Officials: Tommy Hansson, MD, PhD, Principal Investigator — Department of Orthopedics, Sahlgrenska Academy at the University of Gothenburg

REFERENCES:
- [Derived] Olaya-Contreras P, Styf J, Arvidsson D, Frennered K, Hansson T. The effect of the stay active advice on physical activity and on the course of acute severe low back pain. BMC Sports Sci Med Rehabil. 2015 Aug 27;7:19. doi: 10.1186/s13102-015-0013-x. eCollection 2015. PMID 26322232